CLINICAL TRIAL: NCT06322082
Title: Pilates Training Combined With Low Intensity Shock Wave Therapy on Post-prostatectomy Stress Incontinence: Randomized Controlled Trial
Brief Title: Pilates Training and Low Intensity Shock Wave Therapy for Post-prostatectomy Stress Incontinence
Acronym: Incontinence
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Khadra Mohamed Ali (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, Khadra Mohamed Ali, assist professor, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1422024
Record Dates: First submitted 2024-02-14; First posted 2024-03-20 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Stress Incontinence, Male
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Exercise Movement Techniques

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pilates and Shock Wave group (Experimental): 30 patients will receive Pilates exercises combined with Low Intensity Extracorporeal Shock Wave Therapy and conventional pelvic floor muscle exercises
  Interventions: Device: The DUOLITH SD1-TOP focused shock wave system (STORZ MEDICAL AG)
- Shock Wave group (Experimental): 30 patients will receive Low Intensity Extracorporeal Shock Wave Therapy and conventional pelvic floor muscle exercises.
  Interventions: Device: The DUOLITH SD1-TOP focused shock wave system (STORZ MEDICAL AG)
- Pilates group (Experimental): 30 patients will receive Pilates exercises and conventional pelvic floor muscle exercises
  Interventions: Device: The DUOLITH SD1-TOP focused shock wave system (STORZ MEDICAL AG)
- control group (Experimental): 30 patients will receive conventional pelvic floor muscle exercises
  Interventions: Device: The DUOLITH SD1-TOP focused shock wave system (STORZ MEDICAL AG)

INTERVENTIONS:
Device: The DUOLITH SD1-TOP focused shock wave system (STORZ MEDICAL AG) — The LiESWT was applied to Pilates and Shock Wave group and Shock Wave group with 0.25 mJ/mm2 of intensity, 3000 pulses of shock, and 3 pulses/s of frequency, applicator was placed on the suprapubic skin area one session in the week for twelve weeks, totaling 12 sessions.
  Pilates exercises were performed to Pilates and Shock Wave group and Pilates group. The sessions of Pilates were applied twice a week for twelve weeks, totaling 24 sessions. The 50 min Pilates sessions were divided into three phases: warm-up, strengthening, and stretching. They also received written orientations to perform three exercises and two of the Pilates session at home every day - Conventional pelvic floor exercises performed for all groups include Kegel exercise, squats, bridging, and squeeze and release exercises. These exercises were performed 3 times per day, lasting for 12 consecutive weeks
  Other Names: Pilates exercises; conventional pelvic floor muscle exercises

SUMMARY:
120 Patients with urinary incontinence following radical prostatectomy would be randomly assigned to either 4 groups all receive conventional pelvic floor muscle exercises plus group A receive Pilates exercises and Low Intensity Extracorporeal Shock Wave Therapy, group B receive Low Intensity Extracorporeal Shock Wave Therapy, group C receive Pilates exercises and group D receive conventional pelvic floor muscle exercises. Assessment at baseline, immediately after the intervention, to evaluate the degree of urinary incontinence and quality of life after three months from treatment.

DETAILED DESCRIPTION:
120 Patients with urinary incontinence following radical prostatectomy would be randomly assigned to either 4 groups all receive conventional pelvic floor muscle exercises plus group A receive Pilates exercises and Low Intensity Extracorporeal Shock Wave Therapy, group B receive Low Intensity Extracorporeal Shock Wave Therapy, group C receive Pilates exercises and group D receive conventional pelvic floor muscle exercises. Assessment at baseline, immediately after the intervention, to evaluate the degree of urinary incontinence by Urodynamic investigation system, Severity index scale and Cytometry and quality of life by The quality of life questionnaire IQOL after three months from treatment.

ELIGIBILITY:
Inclusion Criteria:

* All patients diagnosed as urinary incontinence.
* Age between 40 -75 male patients or older.
* All patients received the same medical treatment

Exclusion Criteria:

* adjuvant or neoadjuvant chemo-radiation therapy.
* severe postoperative complications.
* history of pelvic surgery, and diseases that could affect voiding function and limitations for the exercise program such as for patients with serious cardiovascular events or spinal or articular disease.

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Cystometry | before treatment and after 3 months
  Ithe dynamic measurement of detrusor pressure during the continuous filling of the bladder.
Severity index scale | before treatment and after 3 months
  measure frequency and amount of urine loss ,calculated by this equation: Severity index of incontinence = (Points for frequency of urine loss) × (Points for amount of urine loss) calculated by this equation: Severity index of incontinence = (Points for frequency of urine loss) × (Points for amount of urine loss) measure frequency and amount of urine loss to calculate severity of incontinence, o Frequency of urine loss grades: Never = 0 less than once a month= 1 once to several times a month = 2 once to several times a week = 3 Every day and/or night = 4
  * o Amount of urine loss grades: No drop (completely dry) = 0 A few drops = 1 A little = 2 More = 3

SECONDARY OUTCOMES:
body mass index | before treatment and after 3 months
  measure ( weight per height squares )of patients kg/m^2

CONTACTS AND LOCATIONS:
Overall Officials: Marwa Eid, Principal Investigator — Professor at Faculty of physical therapy, Cairo University
Locations (1):
- faculty of physical therapy , Cairo university, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes
120 male Patients with urinary incontinence would be randomly assigned to 4 groups all receive conventional pelvic floor exercises(CPFE) plus group A receive Pilates exercises and Low Intensity Extracorporeal Shock Wave Therapy (LiECSWT), group B receive (LiECSWT), group C receive Pilates exercises and group D receive conventional pelvic floor muscle exercises only. (LiECSWT) was applied with 0.25 mJ/mm2 of intensity, 3000 pulses of shock, and 3 pulses/s of frequency, one session in the week for twelve weeks. Pilates exercises twice a week for twelve weeks, totaling 24 sessions and (CPFE) were performed 3 times per day, lasting for 12 consecutive weeks. Assessment at baseline, immediately after the intervention, by Urodynamic investigation system, Severity index scale, Cytometry and The quality of life questionnaire IQOL.
Supporting Information: Study Protocol, ICF
Time Frame: 3 months
Access Criteria: Inclusion criteria :
  * All patients diagnosed as urinary incontinence.
  * Age between 40 -75 male patients or older. • All patients received the same medical treatment
  Exclusion criteria:
  * adjuvant or neoadjuvant chemo-radiation therapy.
  * severe postoperative complications.
  * history of pelvic surgery, and serious cardiovascular events or spinal or articular disease.